CLINICAL TRIAL: NCT04530604
Title: Defibrotide Therapy for SARS-CoV2 Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Defibrotide Therapy for SARS-CoV2 (COVID-19) Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gregory Yanik (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Gregory Yanik, Professor of Pediatric Hematology/Oncology, Professor of Pediatrics and Communicable Diseases and Professor of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00182089
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-06

CONDITIONS: COVID; Sars-CoV2; COVID-19; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — defibrotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Defibrotide (Experimental)
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — All patients will receive 25 milligram/kilogram/day (mg/kg/day) of defibrotide, given in 4 divided doses (approximately every 6 hours), each dose infused over 2-hours intravenously (IV).
  The planned duration of study therapy is 7 days (while in the hospital), with the following qualifications:
  * Patients who respond to study therapy prior to day 7 (able to discontinue oxygen) will discontinue study therapy at that earlier time point.
  * Patients who have not responded to study therapy by day 7 of therapy, evidenced by <20% reduction (or a worsening) of the amount of supplemental oxygen they are receiving, will discontinue study therapy at day 7.
  * Patients who have evidence of a partial pulmonary response by day 7 (>20% reduction in supplemental oxygen requirement, but still require supplemental oxygen) may elect to continue to receive study drug through an additional 7 days of study (total 14-day therapy course).
  Other Names: defitelio

SUMMARY:
This clinical trial will enroll participants that have pneumonia caused by the COVID-19 virus. During the study patients will receive 7 to up to 14 days of defibrotide. After completing the treatment, participants will have 30 day follow-up check-up to assess for adverse events and clinical status. This final assessment can be done virtually, by telephone or electronically (email) if the patient cannot be contacted by phone. No in-person visit is required.

The hypothesis of this trial is that defibrotide therapy given to patients with severe SARS-CoV2 ARDS will be safe and associated with improved overall survival, within 28 days of therapy initiation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of SARS-CoV2 infection, confirmed by real-time reverse transcription polymerase chain reaction (RT-PCR) assay from a nasopharyngeal swab specimen or other diagnostic test for SARS-CoV2.
* Serum D-Dimer ≥ 2.0 mcg/ml.
* Patients with Acute Respiratory Distress Syndrome (ARDS) as determined by the following criteria (Berlin criteria adaptation):

  * Radiographic evidence of bilateral lung disease (opacities or ground glass opacification) on chest radiograph (CXR) or computed tomography (CT), and the opacities not fully explained by pleural effusions, cardiac failure or fluid overload.
  * Impairment of oxygenation, as defined by the ratio of arterial oxygen tension to fraction of inspired oxygen (PaO2/FiO2) ≤ 300 mmHg (millimeters of mercury).
* Patients must provide voluntary written informed consent to be eligible for study. For patients who are medically unable to provide consent, their designated proxy or legal guardian will provide informed consent. The consenting process is described in Appendix II.
* Patients actively participating in another clinical trial for the management of SARS-CoV2 are eligible provided those trials do not directly involve an anti-platelet, anti-coagulant or anti-fibrinolytic agent. (Patients enrolled on investigational trials utilizing anti-viral specific agents, cytokine inhibitors, tyrosine kinase inhibitors, or other anti-inflammatory agents are still eligible).

Exclusion Criteria:

* Concomitant use of heparin, systemic anticoagulants, and/or fibrinolytics are not permitted within 12 hours, with the exception of heparin flushes for centrally placed catheters, fibrinolytic instillation for central venous line occlusion, or in the in-flow circuit for patients on continuous veno-venous hemodialysis.
* Clinically significant acute bleeding, including (but not limited to one of the following): pulmonary hemorrhage (diffuse alveolar hemorrhage), intracranial bleed, gastro-intestinal hemorrhage (gross hematemesis or hematochezia), gross hematuria or uncontrolled epistaxis irrespective of the amount of blood loss, within the prior 3 days.
* On mechanical ventilation for > 96 consecutive hours.
* Serum platelet count < 50,000/Microliters (uL). Transfusion of platelets to achieve a level > 50,000/uL is not allowed for eligibility.
* Serum fibrinogen < 150 mg/dl. Transfusion of fresh frozen plasma or cryoprecipitate to achieve a level > 150 mg/dl is not allowed for eligibility.
* Positive blood culture for a bacterial pathogen within the prior 24 hours prior to study entry, and/or the presence of bacterial pneumonia.
* Hemodynamic instability as defined by a requirement for 2 or more vasopressors (not including renal-doses of dopamine).
* Concurrent use of Extracorporeal membrane oxygenation (ECMO).
* Patients with a previously known hypersensitivity reaction to defibrotide, or any of its excipients.
* Females who are pregnant or breastfeeding.
* History of cerebrovascular accident (i.e. thrombotic or hemorrhagic stroke) within 3 months prior to study entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Yanik, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frame D, Scappaticci GB, Braun TM, Maliarik M, Sisson TH, Pipe SW, Lawrence DA, Richardson PG, Holinstat M, Hyzy RC, Kaul DR, Gregg KS, Lama VN, Yanik GA. Defibrotide Therapy for SARS-CoV-2 ARDS. Chest. 2022 Aug;162(2):346-355. doi: 10.1016/j.chest.2022.03.046. Epub 2022 Apr 9. PMID 35413279

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 13 enrolled, 1 participant was screen failed and did not receive any defibrotide.
Groups:
- Defibrotide: Defibrotide: All patients received 25 milligram/kilogram/day (mg/kg/day) of defibrotide, given in 4 divided doses (approximately every 6 hours), each dose infused over 2-hours intravenously (IV).
  The planned duration of study therapy was 7 days (while in the hospital), with the following qualifications:
  * Patients who responded to study therapy prior to day 7 (able to discontinue oxygen) discontinued study therapy at that earlier time point.
  * Patients who did not respond to study therapy by day 7 of therapy, evidenced by <20% reduction (or a worsening) of the amount of supplemental oxygen they were receiving, discontinued study therapy at day 7.
  * Patients who had evidence of a partial pulmonary response by day 7 (>20% reduction in supplemental oxygen requirement, but still requiring supplemental oxygen) could elect to continue to receive study drug through an additional 7 days of study (total 14-day therapy course).
Period: Overall Study
Arm/Group | Defibrotide
Started | 12
Completed Dosing (One participant discontinued defibrotide early when a pre-therapy blood culture became positive for potential pathogen while the participant was on study therapy. The patient discontinued study at that time but was still evaluable for toxicity and response. Another stopped defibrotide when endotracheal aspirate grew oral flora and H. influenza.) | 10
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Defibrotide
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 0
  30-39 years | 2
  40-49 years | 1
  50-59 years | 2
  60-69 years | 4
  70-79 years | 3
  >80 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Prior Therapy [Count of Participants; unit: Participants]
  Dexamethasone and remdesivir | 9
  Dexamethasone and remdesivir and tocilizumab | 3
Pressors [Count of Participants; unit: Participants] — indicates requirements for vasopressor support at study entry
  Participants | 6
WHO Ordinal Score at Study Entry [Count of Participants; unit: Participants] — Clinical Status Activity and Respiratory Support WHO Ordinal Scores
  1. = Ambulatory, no limitation of activities;
  2. = Ambulatory, Activity LImited;
  3. = Hospitalized, no oxygen therapy;
  4. = Oxygen by mask or nasal cannula;
  5. = Non-invasive ventilation or high-flow oxygen (O2);
  6. = Intubation/mechanical ventilation;
  7. = Intubation/Mechanical ventilation plus one of the following: Pressors, Extracorporeal membrane oxygenation (ECMO) or Dialysis;
  8. = Decased/Death
  Participants
    WHO score of 4 | 2
    WHO score of 6 | 4
    WHO score of 7 | 6
Onset (time in days from diagnosis of SARS - CoV2 to onset of study therapy [Median (Full Range); unit: days] | 9 [1 to 26]
FiO2 [Median (Full Range); unit: Percent] | 55 [40 to 75]
D-dimer (mcg/ml) [Median (Full Range); unit: mcg/ml] | 3.25 [1.33 to 12.3]
Platelets (K/microliter) [Median (Full Range); unit: (K/microliter)] | 226 [70 to 341]
O2 support [Count of Participants; unit: Participants]
  mechanical ventilation | 10
  nasal cannula/ mask | 2
PaO2/FiO2 [Median (Full Range); unit: mmHg] | 137 [83 to 200]
anticoagulant used [Count of Participants; unit: Participants]
  None | 9
  Low Molecular weight Heparin | 2
  Heparin | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Major Hemorrhagic Complications Within 14 Days of Initiation of Treatment
Description: Major hemorrhagic complications will be based on the International Society on Thrombosis and Haemostasis Bleeding scale.
  1. Fatal Bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding associated with a decline in hemoglobin level of > 2.0 g/dl, leading to transfusion of two or more units of whole blood or red cells.
  4. In addition, symptomatic alveolar hemorrhage, macroscopic hematuria, uncontrolled menorrhagia or epistaxis or bleeding from any wound site would also be considered a major hemorrhagic event.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Overall Survival
Description: Number of patients who are alive at Day 28 after starting treatment.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide
Number analyzed (Participants) | 12
Participants | 10

3. Secondary Outcome: Overall Survival
Description: Number of patients who are alive at Day 14 after starting treatment.
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Defibrotide
Number analyzed (Participants) | 12
participants | 11

4. Secondary Outcome: Ventilator-free Survival
Description: Day 14 ventilator-free survival will be summarized by the number of patients who are both alive and not using a ventilator at Day 14 after starting treatment.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide
Number analyzed (Participants) | 12
Participants | 5

5. Secondary Outcome: Number of Ventilator Free Days Within 14 Days of Study Entry
Time Frame: 14 days
Measure: Median (Full Range); unit: days
Arm/Group | Defibrotide
Number analyzed (Participants) | 12
days | 0 [0 to 14]

6. Secondary Outcome: The Time to Improvement in Oxygenation
Description: Improvement in oxygenation defined as an increase in ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) of 50 (or greater) compared to the nadir of PaO2/FiO2.
Time Frame: up to 14 days
Population: 4 participants had improvement by day 14
Measure: Mean (Full Range); unit: days
Arm/Group | Defibrotide
Number analyzed (Participants) | 4
days | 4 [2 to 6]

7. Secondary Outcome: Mean Change in the WHO COVID-19 Ordinal Scale During Therapy
Description: Ordinal scale:
  1. = Ambulatory, no limitation of activities;
  2. = Ambulatory, Activity LImited;
  3. = Hospitalized, no oxygen therapy;
  4. = Oxygen by mask or nasal cannula;
  5. = Non-invasive ventilation or high-flow oxygen (O2);
  6. = Intubation/mechanical ventilation;
  7. = Intubation/Mechanical ventilation plus one of the following: Pressors, Extracorporeal membrane oxygenation (ECMO) or Dialysis;
  8. = Decased/Death Key: For change in ordinal score, negative values represent a decline in WHO score from baseline to day 14 (improvement of condition); positive values represent an increase (worsening of condition).
Time Frame: up to 14 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Defibrotide
Number analyzed (Participants) | 12
score on a scale | -1 [-5 to 1]

ADVERSE EVENTS:
Time Frame: For death and SAEs, participants were followed up at 30 days after completion of therapy; for most participants, 37 days up to a maximum of 44 days. The "other adverse events" table includes any AE (grade 1-5) that occurred during receipt of study drug therapy. Data was collected only during study treatment (7 days for most participants; 14 days for 1).
Description: Participants were already hospitalized and extremely sick so SAEs or AEs after treatment was completed are noted by footnote.
  AEs present at baseline were not recorded as AE, provided there was no clinical worsening of the event during study therapy. Of the 10 out of 12 patients with baseline grade 4 respiratory toxicity, all received mechanical ventilation, and 3 had subsequent progression of respiratory disease and died from progressive respiratory failure after completing study therapy.
Arm/Group | Defibrotide
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide (N=12)
Pulmonary Bacterial Infection (Infections and infestations) | 4 — during treatment
ECMO (Surgical and medical procedures) | 1 — during treatment
Arrhythmia (Cardiac disorders) | 1 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
bleeding/ hemorraghic (Cardiac disorders) | 2 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
Pulmonary fungal infection (Infections and infestations) | 1 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
Pulmonary Bacterial infection (Infections and infestations) | 2 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
Bacterial Infections (Other) (Infections and infestations) | 3 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
Neurologic (Other) (Nervous system disorders) | 1 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
Skin (rash) (Skin and subcutaneous tissue disorders) | 1 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
Tracheostomy (Surgical and medical procedures) | 2 — did not occur during treatment, but occurred within 30 days following completion of defibrotide therapy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide (N=12)
Anemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 3
Thrombocytosis (Cardiac disorders) | 3
Pulmonary Infections (bacterial) (Infections and infestations) | 4
Hypernatremia (Investigations) | 3
Hyperkalemia (Investigations) | 1
Hypercalcemia (Investigations) | 1
Increased ALT (Investigations) | 3
Increased AST (Investigations) | 3
Uremia (Investigations) | 3
alkalosis (Investigations) | 1
creatinine (Renal and urinary disorders) | 1
ECMO (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT04530604/Prot_SAP_000.pdf